CLINICAL TRIAL: NCT00428298
Title: A Double Blind Placebo Controlled Study of Valacyclovir in Cognitive Impairment and Mood Symptoms of Bipolar Disorder
Brief Title: Research Study of Bipolar Mood Symptoms and Cognitive Problems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00009034
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Cognitive; Attention; Memory; Manic Depression; Bi-polar
MeSH Terms: conditions — Bipolar Disorder | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Valacyclovir (Experimental): Subjects dispensed 500 mg capsules. Subjects take two 500 mg capsules twice daily for 16 weeks.
  Interventions: Drug: Valacyclovir
- Placebo Treatment (Placebo Comparator): Subjects dispensed 500 mg capsules. Subjects take two 500 mg capsules twice daily for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Subjects take two 500 mg capsules twice daily for 16 weeks.
  Other Names: Valtrex
  Arms: Active Treatment Valacyclovir
Drug: Placebo — Subjects take two 500 mg capsules twice daily for 16 weeks.
  Arms: Placebo Treatment

SUMMARY:
This is a sixteen week, randomized, double-blind add-on study of valacyclovir versus placebo in approximately 60 outpatients meeting diagnostic criteria according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV Bipolar I or II disorder, testing positive for HSV-1 and who have demonstrable cognitive impairment defined as a total score of less than 85 (one standard deviation from the normal range) on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Each patient will be randomized to double-blind treatment with either valacyclovir or placebo for sixteen weeks. All subjects will be maintained on a stable regimen of psychiatric drugs prescribed by their treating psychiatrist. Patients will be evaluated every 2 weeks by the treatment team and mood rating scales will be administered at each visit including the Young Mania Rating Scale (YMRS) and the Montgomery Asberg Depression Rating Scale (MADRS). The RBANS will be administered again at 8 and 16 weeks. Both the treatment team and the patient will remain blinded during the course of the study. Following the active treatment phase, patients will receive treatment as clinically indicated.

Primary Hypothesis:

Valacyclovir will be superior to placebo in reducing cognitive symptoms associated with bipolar disorder in subjects who have been previously infected with Herpes Simplex virus I (HSV-1).

Secondary Hypothesis:

Valacyclovir will be superior to placebo in reducing mood symptoms associated with bipolar disorder in subjects who have been previously infected with HSV-1.

DETAILED DESCRIPTION:
Background

Herpes Viral Infections and Mental Illness. Recent studies have suggested that chronic, recurrent infections with the herpes family of viruses may play a role in chronic mental illnesses such as schizophrenia and bipolar disorder. Several studies have indicated that individuals with schizophrenia have evidence of increased exposure to Herpes virusesthough this has not been found in all studies . Leweke et al found that untreated individuals with recent first episode schizophrenia had increased levels of serum and cerebrospinal fluid (CSF) immunogloublin G (IgG) antibodies to Cytomegalovirus (CMV) and Toxoplasma gondii in comparison to controls without psychiatric illness. Notably, serum immunoglobulin M (IgM) levels were not increased indicating that infection had not occurred recently. Treated individuals with schizophrenia had similar antibody levels as controls. Finally, Dickerson et al have recently shown that previous Herpes Simplex Virus -1 (HSV-1) infection is associated with cognitive impairment in bipolar disorder, with a relative risk of 22.2 and that this risk was increased in the presence of the catechol-o-methyltransferase (COMT) 158 Val/Val genotype.

It is well known that active replication of herpes viruses may occur after extended periods of latency. It has also been shown active replication of the virus in the central nervous system may be triggered by environmental or psychosocial stressors and cause mood and even psychotic symptoms. Taken together with the evidence of increased exposure to Herpes viruses found in individuals with schizophrenia and bipolar disorder, one hypotheses that remains to be tested is that episodic reactivation of Herpes Simplex 1 (HSV-1) in the brain triggered by environmental stressors could be a pathogenic mechanism contributing to symptomatology in a subset of bipolar disorder and schizophrenic patients.

Cognitive Impairment in Bipolar Disorder

Cognitive, or neuropsychological, functioning is one of the major domains of symptomatology in major mental illness. While cognitive impairment in schizophrenia has been long established, neuropsychological functioning in bipolar disorder has been less extensively studied. Nevertheless, there is evidence that patients with mood disorders frequently manifest cognitive deficits in attention, executive and memory functions. While symptomatic bipolar disorder patients have been shown to have widespread cognitive abnormalities, evidence from many studies also supports the hypothesis that there are persistent residual cognitive impairments in patients in the euthymic phase of illness. As noted above, Dickerson et al have very recently shown an association between HSV-1 seropositivity and cognitive dysfunction in bipolar disorder (2006).

Valacyclovir in Schizophrenia

Recent studies have shown that herpes viruses may play an etiologic role in the cognitive impairments that occur in a subset of patients with schizophrenia and bipolar disorder. Dickerson et al. found that serum antibodies to HSV1 were an independent predictor of cognitive dysfunction in schizophrenia. Similarly, Dickerson et al. found that serological evidence of infection with HSV1 was also predictive of cognitive impairment in bipolar disorder. This association was independent of other factors that could affect cognition including manic, depressive and psychotic symptoms, age of onset, education, or medications. A clinical trial using the antiviral medication valacyclovir in schizophrenia was recently conducted. This study found a significant improvement in psychiatric symptoms in individuals with schizophrenia who were seropositive for cytomegalovirus, another virus in the herpes family. This is the first evidence that an antiviral medication may be helpful in a psychiatric condition.

The study will be divided into two phases

Screening Phase. Subjects will initially be screened by telephone and, if they meet major inclusion and exclusion criteria, will then be invited for an in-person screening. After a consenting process, subjects will first under go RBANS testing. If they meet criteria for cognitive impairment (total score <85) subjects will then go one to have a rapid HSV1 test administered (result available in 1-7 days at Hopkins) and will undergo the Structured Clinical Interview for the Diagnostic and Statistical Manual IV (SCID) conducted by a research assistant. Subjects who test positive for HSV-1 and who have a diagnosis of Bipolar I or Bipolar II disorder on the SCID will be invited back to meet with a team psychiatrist to complete the screening, including a psychiatric interview and examination, a medical history and physical examination, vital signs, and baseline laboratory tests including a complete blood count and blood chemistries as well as any other evaluation the treatment team feels is medically indicated. Subjects who are appropriate for the study will be invited to join the Active Phase of the study.

Active Phase

A second consenting process will be conducted for entrance into the active phase of the trial. Subjects will enter this phase within 14 days of the RBANS testing of the screening visit. During this phase the patients will be randomly assigned to receive either valacyclovir or placebo in addition to their standard psychiatric medications. The patients will receive capsules containing valacyclovir or placebo and will be blinded during the course of the study. Valacyclovir will be started at a initial dose of 1000mg twice daily. At the baseline visit, mood rating scales including the YMRS, MADRS, and PANSS will be administered. Subjects will then meet with the treatment team every 2 weeks for rating scale measurements and assessments for side effects. At the end of 8 and 16 weeks, subjects will again undergo RBANS testing. Both subjects and raters will remain blind during the trial

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Have a diagnosis of Bipolar I or II disorder (as defined by DSM-IV)
* Be in active treatment with an outpatient psychiatrist
* Test positive for HSV1
* Demonstrate cognitive impairment on the RBANS as defined by a total score of less than 85 (i.e. greater than one standard deviation below normal).

Exclusion Criteria:

* Either pregnant or nursing
* Have been diagnosed with any serious, unstable illnesses including HIV infection or other immunodeficiency condition, hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease and hypertension), endocrinologic, neurologic, immunologic, or hematologic disease. Illnesses that are currently well controlled and being treated are not grounds for exclusion.
* Have a history of hypersensitivity or intolerance to valacyclovir or acyclovir
* Meet criteria for DSM-IV substance abuse (except nicotine and caffeine) within the past 90 days
* Had Electroconvulsive Therapy (ECT) within three months prior to randomization
* Judged to be at serious suicidal risk; inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Payne, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Dept. of Psychiatry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickerson FB, Boronow JJ, Stallings CR, Origoni AE, Yolken RH. Reduction of symptoms by valacyclovir in cytomegalovirus-seropositive individuals with schizophrenia. Am J Psychiatry. 2003 Dec;160(12):2234-6. doi: 10.1176/appi.ajp.160.12.2234. PMID 14638597
- [Background] Dickerson FB, Boronow JJ, Stallings C, Origoni AE, Cole S, Krivogorsky B, Yolken RH. Infection with herpes simplex virus type 1 is associated with cognitive deficits in bipolar disorder. Biol Psychiatry. 2004 Mar 15;55(6):588-93. doi: 10.1016/j.biopsych.2003.10.008. PMID 15013827
- [Background] Dickerson FB, Boronow JJ, Stallings C, Origoni AE, Sullens A, Yolken RH. The catechol O-methyltransferase Val158Met polymorphism is not associated with broad-based cognitive functioning in schizophrenia. Schizophr Res. 2007 Nov;96(1-3):87-92. doi: 10.1016/j.schres.2007.05.021. Epub 2007 Jul 2. PMID 17601704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment Valacyclovir | Placebo Treatment
Started | 30 | 30
Second RBANS at Study Exit | 3 | 3
Completed | 16 | 19
Not Completed | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Valacyclovir | Placebo Treatment | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (7) | 41 (10) | 42 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status at 16 Weeks
Description: The RBANS is a brief, independently administered measurement of cognitive decline or improvement.
  The test is comprised of 12 subtests which comprise 5 domains. The age of the participant and the scores from each domain inform the total RBANS score (Index Score) analyzed in this study. The range for total score is 40-160. If the total score for a subject increases this denotes improved performance on the RBANS.
  The RBANS was administered at baseline and 16 weeks.
Time Frame: 16 weeks
Population: Participants who completed screening/first visit Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and study completion/last visit RBANS. Discrepancies in number of participants analyzed are due to subjects who dropped out and did not have final RBANS scores. Imputed data was used for those participants.
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Active Treatment Valacyclovir | Placebo Treatment
Number analyzed (Participants) | 19 | 22
percentage of change | 10.1053 [2.074 to 18.1366] | 3.6364 [-.05218 to 7.7946]

2. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Score at 16 Weeks
Description: The MADRS is a 10 item depression rating scale administered by a research team member. The MADRS is composed of 10 items with a 7 point fixed rating scale (0-6). A higher score indicates the presence of depressive symptoms.
Time Frame: 16 weeks
Population: Discrepancies in number of participants analyzed are due to subjects who dropped out and did not have final assessments. Imputed data was used for those participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Treatment Group - Valcyclovir; Inactive Treatment Group - Placebo: Subjects dispensed 500 mg capsules. Subjects take two 500 mg capsules twice daily for 16 weeks.
Arm/Group | Active Treatment Group - Valcyclovir | Inactive Treatment Group - Placebo
Number analyzed (Participants) | 19 | 22
units on a scale
  Baseline MADRS | 27.94 (11.73) | 19.74 (12.09)
  Final MADRS 16 weeks | 11.5 (9.76) | 14.89 (13.17)

3. Other Pre Specified Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) at 16 Weeks
Description: The Young Mania Rating Scale has 11 items that rate the subject's subjective experience and clinician observation. Four items are rated 0-8, the remaining are rated 0-4.
  The score can range from 0 to 60. A higher score indicates the presence of manic symptoms.
Time Frame: 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment Group - Valcyclovir | Inactive Treatment Group - Placebo
Number analyzed (Participants) | 19 | 22
units on a scale
  Baseline YMRS | 7.88 (5.84) | 8.84 (8.08)
  Final YMRS 16 weeks | 5.19 (5.67) | 4.84 (5.18)

ADVERSE EVENTS:
Arm/Group | Active Treatment Valacyclovir | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No